CLINICAL TRIAL: NCT00029289
Title: Effects of Lutein in Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000292-01 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Lutein

INTERVENTIONS:
Drug: Lutein (10 or 30 mg/day) capsules

SUMMARY:
Phase I/II double-masked, randomized, placebo-controlled, cross-over trial to determine effects of lutein on vision in retinitis pigmentosa, including safety and effective dosage assessment

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a group of congenital retinal degenerations affecting over 100,000 individuals in the US, characterized by nightblindness, gradual loss of peripheral vision, and eventually total vision loss. Despite surgical and medical efforts it has not been possible to slow down, let alone reverse, the process of photoreceptor degeneration in RP. However, a recent patient-initiated pilot study demonstrated that RP patients may respond to a nutrition supplement (lutein) with a modest, but statistically significant gain in visual acuity and central visual field area; demonstration of these effects relied critically on frequent home vision tests using a letter chart on the screen of a personal computer and a wall chart to measure the central visual field. Supporting the reliability of the data was a highly significant correlation between eye color and vision changes; eye color has earlier been shown to influence macular pigment changes following lutein supplementation.

At this state, a study of long-term lutein benefits would be costly and, without placebo-controlled pilot data, premature. We are proposing to prepare for a long-term clinical trial through an exploratory study, investigating the effects of lutein and creating PC-based home vision tests. In the initial 6 months of the study, we will develop and adapt standard clinical vision tests for use on a personal computer, and recruit two study groups: 1) 42 RP patients to study the effects of lutein on vision, using placebo and 20 dosages in a randomized, double-masked crossover design (Latin Square, 2x16 weeks), testing for possible adverse effects through serum hepatic panels every 4-6 weeks, and measuring compliance through baseline and end-value serum carotenoid tests and frequent macular pigment density tests; 2) 31 other volunteers (10 normally signed, 21 RP patients) who, along with the first group, will monitor their vision every 1-2 weeks at home using the PC-based tests. Results will be validated against those obtained with standards tests during multiple visits to our center.

The results and tools produced by this study will enable a long-term lutein supplementation trial with vision as its principal outcome measure, and the study can serve as a model for other supplement trials. Moreover, by virtue of the PC-based home vision tests developed as part of this study, such future trials may, under proper safeguards, enroll remote participants who would download test software, perform frequent outcome tests at home, submit test results via e-mail, and be examined periodically by local physicians to detect potential adverse effects.

Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Wilmer Eye Institute, Lions Vision Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bahrami H, Melia M, Dagnelie G. Lutein supplementation in retinitis pigmentosa: PC-based vision assessment in a randomized double-masked placebo-controlled clinical trial [NCT00029289]. BMC Ophthalmol. 2006 Jun 7;6:23. doi: 10.1186/1471-2415-6-23. PMID 16759390